CLINICAL TRIAL: NCT05056194
Title: A Double-blind, Randomized, Placebo-controlled, Parallel, Study to Assess the Efficacy and Safety of XW10172 MR for the Treatment of Excessive Daytime Sleepiness in Patients with Parkinson's Disease
Brief Title: Valiloxybate (XW10172 MR) Efficacy and Safety Parkinson's Disease Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: XWPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XW10172-104
Record Dates: First submitted 2021-09-17; First posted 2021-09-24 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease; Excessive Daytime Somnolence
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valiloxybate (Experimental): XW10172 Modified Release (MR) Granules for Oral Suspension
  Interventions: Drug: Valiloxybate
- Placebo (Placebo Comparator): Placebo Granules for Oral Suspension
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Valiloxybate — XW10172 MR Granules for Oral Suspension
  Other Names: XW10172 MR
  Arms: Valiloxybate
Other: Placebo — Placebo Granules for Oral Suspension
  Arms: Placebo

SUMMARY:
Following screening visit and verification of inclusion/exclusion criteria and informed consent, participants will undergo a multiple sleep latency test (MSLT) and polysomnogram (PSG) assessments to confirm eligibility for randomization. Participants will be randomized to two groups: placebo or XW10172 MR. The drug will be taken orally at bedtime for 6 weeks of treatment that will consist of a 2-week dose escalation/titration period and a 4-week stable-dose maintenance period. There will be a 2-week safety period following dosing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease consistent with the UK-PD Society Brain Bank Criteria and PD duration at least 1 year with modified Hoehn and Yahr stage 1-3 in the OFF state.
* Patient reported history of excessive daytime sleepiness (e.g., frequent dozing, nodding, or naps).
* Anti-Parkinson's medications at stable doses for at least 1 month prior to the Baseline Visit and can maintain a fixed, stable dose throughout the study
* Epworth Sleepiness Scale score of >10 at screening.
* Female participants of childbearing potential must test negative in a serum pregnancy test at Screening and have a negative urine pregnancy test at the Baseline and Visit. Women with childbearing potential must use an acceptable method of contraception during the study and for at least 30 days after completion of dosing.

Exclusion Criteria:

* Atypical or secondary parkinsonism
* Significant medical conditions.
* Evidence of moderate or severe sleep disordered breathing.
* Drugs that affect sleep including CNS depressants and stimulants.
* Montreal Cognitive Assessment (MoCA) examine score <24.
* Hospital Anxiety and Depression Scales (HADS) >11.
* Have an occupation that requires variable shift work or routine night shifts or travel across two or more-time zones.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Difference between XW10172 MR and placebo in the change from baseline to end-of-maintenance in the Epworth Sleepiness Scale. | 6 weeks

SECONDARY OUTCOMES:
Difference between XW10172 and placebo in the change from baseline to end-of-maintenance in the Caregiver Global Impression of Change. | 6 weeks
Difference between XW10172 MR and placebo in the change from baseline to end-of-maintenance in the Multiple Sleep Latency Test | 6 weeks
Difference between XW10172 MR and placebo in the change from baseline to end-of-maintenance in the Parkinson's Fatigue Scale 16. | 6 weeks
Difference between XW10172 MR and placebo in the change from baseline to end-of-maintenance in the Brief Assessment of Cognition composite score | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Canafax, PharmD, Study Director — XWPharma

IPD SHARING:
Plan to Share IPD: No